CLINICAL TRIAL: NCT07067021
Title: Detection of Postoperative Gastrointestinal System Dysfunctions in Patients Undergoing Cesarean Section With Transabdominal Block Under General Anesthesia"
Brief Title: Post-Cesarean Gastrointestinal Dysfunction
Status: Completed | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Sponsor
Other Study IDs: FSCH-SB-2024/06-15
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Cesarean Section Surgery; TAP Blocks; Gastrointestinal Dysfunction
Keywords: Cesarean Section; TAP Block; Gastrointestinal Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group T: Patients who received a TAP block under general anesthesia.: Group T: This group consists of patients who underwent Cesarean section under general anesthesia and received a Transabdominal Plane (TAP) block during the surgery. The TAP block is a regional anesthetic technique administered for postoperative pain management.
- Group C: Patients who did not receive a TAP block.: Group C (Control Group) Description: This group consists of patients who underwent Cesarean section under general anesthesia but did not receive a TAP block during the surgery. This group will receive standard postoperative pain management for comparison with the effects of the TAP block.

SUMMARY:
General anesthesia has a range of effects that can lead to gastrointestinal (GI) system dysfunctions in the postoperative period. These effects are linked to various factors, from the pharmacological properties of anesthetic agents to neurohumoral effects triggered by surgical stress. Commonly encountered GI dysfunctions include nausea and vomiting, abdominal distension due to decreased intestinal peristalsis and the postoperative inflammatory response, delayed gastric emptying, ileus, fatigue, and delayed initiation of oral feeding. These conditions can prolong hospital stay, increase treatment costs, and reduce patient comfort.

In clinical practice, protecting GI function and preventing complications after general anesthesia are of great importance. One of the main goals of applying Enhanced Recovery After Surgery (ERAS) protocols is to reduce the surgical stress response, thereby promoting rapid recovery and improving GI functions.

Postoperative gastrointestinal (GI) dysfunction after cesarean section is a common complication that negatively impacts the recovery process. This condition manifests with symptoms such as abdominal pain, nausea, vomiting, and an inability to pass flatus, and it can prolong hospital stay and increase costs. Opioid analgesics are known to negatively affect postoperative GI motility, and regional anesthesia techniques can alleviate these problems by reducing opioid requirements. Fascial plane blocks like the TAP block are thought to reduce somatic and visceral pain by injecting local anesthetics between the deep and superficial layers of the fascia, and may positively influence GI functions through sympathetic blockade.

This study aims to observationally investigate the effect of ultrasound-guided transabdominal plane (TAP) block on postoperative gastrointestinal system (GI) dysfunctions in patients who have undergone cesarean section.

DETAILED DESCRIPTION:
Postoperative Gastrointestinal Dysfunction (POGD) refers to a collection of clinical symptoms that arise after general anesthesia, encompassing disruptions in normal gastrointestinal (GI) peristaltic activity and imbalances in absorption and secretion. This condition develops as a result of a complex interaction of neurological, inflammatory, pharmacological, and metabolic factors. These symptoms include nausea and vomiting, gastroparesis, delayed flatus and defecation, delayed oral feeding, abdominal distension, and pathophysiological changes like paralytic ileus.

Many risk factors affect POGD after Cesarean Delivery (CD) surgery. Predisposing factors include the surgical method, degree of abdominal adhesions, amount of opioid use, postoperative blood transfusion, bowel manipulation, duration of surgery, advanced age, and infection and inflammation statuses.

In patients undergoing CD under general anesthesia, POGD disorders are observed due to surgical stress and opioid use. The Enhanced Recovery After Cesarean Delivery (ERAC) protocol offers a multidisciplinary, holistic approach that reduces POGD and accelerates maternal recovery through a set of perioperative care guidelines.

The Transabdominal Plane (TAP) block, a regional anesthesia technique with proven efficacy in postoperative pain management after CD, holds an important place within the modern multimodal analgesia approach of ERAC protocols. By reducing opioid consumption, it decreases the prevalence of POGD and enhances maternal comfort, indirectly contributing to newborn care.

To reflect patients' subjective experiences regarding postoperative GI symptoms, the PRO-diGI (Patient-Reported Outcome Measure for Gastrointestinal Dysfunction after major abdominal surgery) scale has been developed and is being effectively used. The Obstetric Quality-of-Recovery score (ObsQoR-11) is a Patient-Reported Outcome Measure (PROM) developed to comprehensively and standardly assess the quality of maternal recovery after childbirth. This score, whose reliability and validity have been proven in the Turkish population (ObsQoR-11T), clinically and objectively evaluates the postpartum period by considering both physical symptoms and the mother's psychological well-being and functional capacity.

This study aims to determine the effects of ultrasound-guided TAP block on recovery quality assessment (ObsQoR-11T score), postoperative gastrointestinal dysfunction (PRO-diGI score), and gastrointestinal motility (Perlas Score determined by USG) in patients who have undergone CD.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cesarean section surgery under general anesthesia

Patients with American Society of Anesthesiologists (ASA) physical status I-II-III

Patients able to understand and respond to the Visual Analog Scale (VAS) for pain

No history of drug or alcohol addiction

No coagulation disorders

No anatomical abnormalities of the gastrointestinal system

No gastrointestinal motility disorders

No previous abdominal surgery

No allergies to local anesthetic drugs

No history of diabetes mellitus

No severe systemic diseases

No intraoperative surgical complications (such as bleeding, conversion to open surgery, or organ injury)

Successful block achievement (for relevant groups)

Exclusion Criteria:

* Patients undergoing emergency cesarean section under general anesthesia

Patients with American Society of Anesthesiologists (ASA) physical status IV-V

Patients unable to understand the Visual Analog Scale (VAS) for pain (due to cognitive or psychiatric disorders, or mental impairments)

Emergency operations

Patients with drug or alcohol addiction

Coagulation disorders

Anatomical abnormalities of the gastrointestinal system

Gastrointestinal motility disorders

Previous abdominal surgery

Allergy to local anesthetic drugs

Diabetes mellitus

Presence of severe systemic disease

Intraoperative surgical complications (such as bleeding, conversion to open surgery, organ injury, etc.)

Unsuccessful block placement

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Turkish kohort
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
PRO-diGI (Patient-Reported Outcome Measure for Gastrointestinal Dysfunction after major abdominal surgery) | 24. hour, 48. hour, 72. hour
  Patients will be asked 15 questions from the PRO-diGI (Patient-Reported Outcome Measure for Gastrointestinal Dysfunction after major abdominal surgery) scale to assess GI dysfunction.The first response option was given the highest score of 4 points, and the last response option was given the lowest score of 0 points. Patients received a maximum score of 60 points when their GI function was in the best condition.

SECONDARY OUTCOMES:
The Obstetric Quality-of-Recovery score (ObsQoR-11) | 24. hour
  The Obstetric Quality-of-Recovery score (ObsQoR-11) is a Patient-Reported Outcome Measure (PROM) developed to provide a standardized and comprehensive assessment of maternal postpartum recovery quality.The ObsQoR-11 score is a scale used to assess the quality of recovery in mothers after a cesarean section, ranging from 0 (indicating the worst recovery) to 110 (indicating the best recovery); higher scores signify a better quality of recovery in terms of the mother's physical symptoms, psychological well-being, and functional capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided